CLINICAL TRIAL: NCT02140853
Title: Multi-drug Resistant Gram-negative Bacilli-surveillance and Clinical Feature in China
Brief Title: MDR Bacilli Surveillance and Clinical Feature in China
Acronym: MDR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Prof Xie Canmao, Director, Respiratory Department, Sun Yat-sen University
Other Study IDs: WS1993136; MDR Net (Other Grant/Funding Number: Pfizer, WI1993136)
Record Dates: First submitted 2014-05-14; First posted 2014-05-16 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Infection
Keywords: MDR gram-negative bacilli; Mortality; Therapy
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — sputum, pleural effusion or blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- MDR group: patients of MDR pathogen infection
- non-MDR group: patients of non-MDR pathogen infection

SUMMARY:
Objective

1. To evaluate the impact of MDR pathogen on prognosis and therapy cost;
2. To compare the efficacy of different antibiotics in treatment of infection caused by MDR pathogens;
3. To evaluate the risk factors of MDR pathogens infection;
4. To evaluate the distribution and characteristics of MDR pathogens;
5. To investigate the proportion of MDR isolates to construct systematic database.

DETAILED DESCRIPTION:
1. Background:

   In recent years, the incidence of infection caused by multi-drug resistant (MDR) pathogen keeps increasing. The increase of MDR bacterial is a serious challenge for empirical therapy. Common empirical antibiotic may not cover MDR pathogen and is inappropriate for patients with infection caused by MDR pathogens, which finally increases mortality. A number of studies have demonstrated MDR pathogens are related to excess mortality, longer hospital stays and more treatment cost. Compared to infection caused by non-MDR pathogens, infection caused by MDR pathogens possesses higher mortality by 10% to 15%, longer ICU stays by 6 -10 days, and less appropriate empirical antibiotics by 50%. In addition, studies have shown that the treatment of infection caused by MDR pathogens is more expensive by $10,000-$50,000 than that by sensitive pathogens. Monitoring of MDR pathogens may find epidemiological trends, discover new MDR bacteria, evaluate risk factors and assess the effectiveness of interventions. Data of MDR pathogens has been available in Europe and the United States, however, is absent in China. By now, the features of bacterial resistance in different regions, hospitals, or in certain patients with exposure to antibiotics, still keep uncertainty.

   The current study is to enroll continuous MDR isolates and clinical data of the patients from which the pathogens were isolated. The data may clarify the distribution and characteristics of MDR pathogens in China, as well as clinical outcome of infection caused by MDR pathogens, which is essential for management and treatment of infection caused by MDR pathogens.
2. Study center: 10
3. Strains MDR gram-negative bacilli isolated from lower respiratory tract, pleural effusion or blood will be reported to clinician. Confirmation that the isolate is 'real' pathogen of a certain infection, not colonization or pollution, is needed. Microbiologic data will be collected, such as result of susceptibility test.

   Inclusion criteria:
   1. Gram-negative bacillus.
   2. Resistant to more than 3 kinds of antibacterial agents.

   Exclusion criteria:
   1. Repetitive organism isolated from the same center in one patient.
   2. Judged as colonization or pollution by clinician.
   3. Enrolled into other trial, and the data is not available for the current study.
4. Microbiologic investigators collect data:

   1. General data, strain name, source department.
   2. Result of susceptibility test.
5. Clinical data:

   The current trial is observational. Clinicians, rather than investigators, will decide the therapy. Clinical investigators confirm the MDR organism is not pollution or colonization by both definitions of nosocomial infection and result of semi-quantitative culture.

   For those eligible strains, corresponding clinical data will be collected.
   1. Demographic data. Name, gender, age and date of admission.
   2. Symptoms and signs, especially those related to infection.
   3. Laboratory result, such as blood and urine routine, biochemistry.
   4. Medical complication, especially those that influence immunity, such as diabetes, hepatic cirrhosis, malnutrition, malignancy, HIV infection or transplantation.
   5. Previous medical therapy, especially late usage of antibiotic, steroids or other immunosuppressive agents.
   6. Management of infection, including regimen and duration of antibiotic therapy, prognosis, treatment and total cost.
   7. Outcome of treatment, including efficacy at the end of antibiotic therapy and 30-day, ICU stay time, total hospital stay, and cost of antibiotic and totaltherapy cost.
6. Sample size:

   Continuous MDR gram-negative bacilli and clinical data: 1500 cases. Continuous Non-MDR gram-negative bacilli and clinical data: 1500 cases.
7. Endpoint:

   1. Mortality and therapy cost of MDR or non-MDR infection.
   2. Success rate of different antibiotics regimen for treatment of MDR infection. (Classified as 3rd and 4th cephalosporin,β-lactam and β-lactamase inhibitor compounds, carbapenems and others, monotherapy or combined therapy)
   3. Risk factors of infection caused by MDR pathogens.
   4. Resistant profile of MDR bacilli responsible for infection.
   5. Therapy cost of MDR or non-MDR infection.
8. Statistical analysis:

Statistical analysis is conducted by t-test for continuous variables and chi-square test for categorical variables. Multivariate regression analysis, Logistic regression model is used to clarify the independent risk factors of infection and death. All p values are retained until after the decimal point two, and statistical significance was set at p <0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Gram-negative bacillus.
2. Resistant to more than 3 kinds of antibacterial agents.

Exclusion Criteria:

1. Repetitive organism isolated from the same center in one patient.
2. Judged as colonization or pollution by clinician.
3. Enrolled into other trial, and the data is not available for the current study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 3000
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2011-11; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | Jun 2015
  Mortality comparizon between MDR or non-MDR infection

SECONDARY OUTCOMES:
Therapy cost | Jun 2015
  Therapy cost comparizon between MDR or non-MDR infection

OTHER OUTCOMES:
Success rate of different antibiotics regimen for treatment of MDR infection | Jun 2015

CONTACTS AND LOCATIONS:
Overall Officials: Canmao Xie, MD, Principal Investigator — Sun Yat-sen University; Yuxing Ni, MD, Principal Investigator — Ruijin Hospital
Locations (1):
- SunYat-senU, Guangzhou, Guangdong, China